CLINICAL TRIAL: NCT06588842
Title: Cluster Set Resistance Training as a Modality of Power Training in Older Adults
Brief Title: Cluster Resistance Training and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240776
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Healthy Aging
Keywords: Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cluster Set Resistance Training (Experimental): Participants in this group will receive high-speed resistance training 2 times a week for 12 consecutive weeks.
  Interventions: Other: Cluster Set Resistance Training
- Traditional Set Resistance Training (Active Comparator): Participants in this group will receive traditional set resistance training 2 times a week for 12 consecutive weeks.
  Interventions: Other: Traditional Set Resistance Training

INTERVENTIONS:
Other: Cluster Set Resistance Training — Participants will receive a total of 24 in-person training sessions using three sets of eight repetitions per set. During training participants will be allowed 1-minute rests between sets and 15-second rests after repetitions three and six.
  Arms: Cluster Set Resistance Training
Other: Traditional Set Resistance Training — Participants will receive a total of 24 in-person training sessions using three sets of eight repetitions per set. During training participants will be allowed 1-minute rests between sets.
  Arms: Traditional Set Resistance Training

SUMMARY:
This project will focus on improving power in older adults, since power is related to performance of daily activities and memory and decision making. The study will compare cluster set resistance training, where you can rest during a set, to traditional set resistance training where all repetitions in a set must be completed without any between-repetition rest. If cluster set resistance training is better than traditional set resistance training, it could be more beneficial than existing methods in improving independence in older persons.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment Score > 23
* No memory complaints

Exclusion Criteria:

* Uncontrolled cardiovascular or neuromuscular disease that prevents participation in a training program
* Any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, system lupus erythematosus, or other serious concomitant medical illness
* Unresolved injury or surgery to the upper or lower limbs.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in neuromuscular performance as measured by power production. | Baseline, 12 weeks
  This test measures the power a person can produce at maximal speed using a load of 50% of 1RM for the chest press and leg press. There are no minimum or maximum scores. The higher score is better. Power shows how fast a person can do work. The test typically takes about five minutes. Unit of measure is Watts.
Change in neuromuscular performance as measured by 1-repetition maximum (1RM) | Baseline, 12 weeks
  Maximal load that can be lifted in one repetition (1RM) will be assessed for in both leg press and chest press exercises. The loads on the testing equipment will be increased over 5 to 7 testing sets. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test.
  The test typically takes 5 to 10 minutes. The higher the 1RM the stronger the person is.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Baseline, 12 weeks
  The MoCA is a brief cognitive screening tool with high sensitivity and specificity for detecting mild cognitive impairment. The MoCA has 16 items. If cognitive impairment is detected through this screening questionnaire, subjects will not be included in the research. The scale has a total score of 30 points. ≥26 points were considered as having no cognitive impairment.
Change in the Hopkins Verbal Learning Test | Baseline, 12 weeks
  The Hopkins Verbal Learning Test is a brief assessment of immediate recall, delayed recall and delayed recognition commonly used with populations with Alzheimer's disease, Huntington's disease and amnesic disorders. The maximum score for the test is 36 with scores below 14, indicating dementia. The minimum score is 0 and the maximum score is 36. A higher score indicates better working memory. The test takes about 5-10 minutes to take.
Change in Concept Switching as measured by the Dimensional Card Sort test. | Baseline, 12 weeks
  The Dimensional Change Card Sort test is a measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). Four trials are also employed, in which the participant must change the dimension being matched. Scoring is based on a combination of accuracy and reaction time. Scores can range from 0-10. The higher the score, the better the capacity to switch from one concept to another. The test typically lasts four minutes.
Change in the Flanker test | Baseline, 12 weeks
  The Flanker Test uses response inhibition to assess a subject's capacity to suppress incorrect responses within a particular context. The target (for this study an arrow) is flanked by non-target arrows that are either in the same direction as the target (congruent flankers), the opposite response (incongruent flankers), or to neither (neutral flankers). The minimum score is 0 and the maximum score is 10. A higher score indicates better accuracy. The test takes about 3 minutes.
Change in Event Memory as measured by the Picture Sequence Memory Test | Baseline, 12 weeks
  The Picture Sequence Memory Test (PSMT) can test how well a subject can remember events. The participants are asked to recall the sequence of pictures presented over two learning trials. Participants are given credit for each adjacent pair of pictures they correctly put in place. The minimum score is 0 and the maximum score is 17. The higher the score indicates better sequential memory. The test takes approximately seven minutes to administer.
Change in Information Sorting as measured by the NIH List Sorting Test | Baseline, 12 weeks
  The National Institute of Health (NIH) List Sorting Test measures a person's ability to store information for a short time while doing other tasks. It asks the subject to sort and put in order lists of both sounds and pictures. The lists may include animals to be sorted by size, foods to be sorted by size, or a combination of the two to be sorted by size. The minimum score is 0 and the maximum score is 26. A higher score indicates better working memory. The test takes about 7 minutes.
Change in Reaction Time for a Mental Task as measured by the NIH Pattern Comparison Processing Speed Test | Baseline, 12 weeks
  The Pattern Comparison test measures the subject's reaction time and how long it takes the subject to do a mental task. During the test, the subject will be asked to decide whether two visual patterns are the same or not the same. The minimum score is 0 and the maximum score is 130. A higher score indicates better processing speed. The test takes 85 seconds.
Change in Mental Task as measured by Trail Making Test | Baseline, 12 weeks
  Used to assess executive function in the areas of visual attention (Part A) and set-shifting (the ability to shift attention between one task and another; Part B). The time to complete this test is recorded in seconds.
Change in the Speed of the Ten-Meter Walk Test | Baseline, 12 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when they cross the 10-m mark. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed, and the average will be documented in meters per second. One-minute recoveries will be provided between trials. Total time is 7 minutes.
Change in Time for the Five Times Sit-to-Stand Test | Baseline, 12 weeks
  The five time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with their arms folded across their chest and their back against the chair. On verbal command, the participant will stand up and sit down 5 times as quickly as possible. Timing begins at "Go" and ends when the buttocks touch the chair after the 5th repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Change in Distance of the Seated Medicine Ball Throw | Baseline, 12 weeks
  For the Seated Medicine Ball Throw, subjects will sit in an armless chair with their back against the chair back, while holding the 6-pound medicine ball against their chest. Subjects will then throw the ball at a perceived 45° angle as far as possible. Subjects must complete at least three practice trials; however, subjects will be allowed more trials until comfortable with the testing procedure. Upon starting the official trial, subjects will complete three separate attempts at each varying medicine ball, to nine trials in total. Each of the three trials within a given medicine ball will be separated by a 1-minute rest. Distance will be measured in centimeters.
Change in the time required to complete the timed Up-and-Go Test. | Baseline, 12 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair, and then returns to a seated position as quickly as possible. Time is measured in seconds. The faster the person completes the test the better the dynamic balance.
Change in Muscle Thickness using Ultrasound | Baseline, 12 weeks
  Three images will be taken in the longitudinal view in B-mode. Muscle thickness will be measured by drawing a perpendicular line from the deep to superficial aponeurosis at the thickest region of each muscle. The unit of measurement is centimeters
Change in Muscle Quality using Ultrasound | Baseline, 12 weeks
  Muscle quality will be measured using a gray scale. The black and white pixels correspond to arbitrary values of 0 (darker) to 255 (lighter), with darker colors indicting more muscle and lighter colors indicating more fat.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No